CLINICAL TRIAL: NCT05087186
Title: Psychological Support for Intensive Care Nurses During the COVID-19 Pandemic: The PROACTIVE Feasibility Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRI0412
Record Dates: First submitted 2021-10-18; First posted 2021-10-21 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Psychological; Burnout; Post Traumatic Stress Disorder; Anxiety; Depression
Keywords: Critical Care; Intensive Care; Staff Wellbeing; Guided Imagery; FLASH technique
MeSH Terms: conditions — Burnout, Psychological; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Group sessions with psychological therapists
  Interventions: Behavioral: Guided imagery and FLASH technique

INTERVENTIONS:
Behavioral: Guided imagery and FLASH technique — Five virtual group sessions delivered by psychological therapists;
  * Sessions 1 and 2: Guided imagery
  * Sessions 3 and 4: FLASH technique
  * Session 5: Refresher on guided imagery and FLASH technique

SUMMARY:
The psychological health of frontline healthcare workers, caring for critically ill patients with COVID-19, has deteriorated during the pandemic. Nurses appear to be most seriously affected. Despite the availability of supportive interventions, uptake is poor, and none have been found beneficial in randomised controlled trials.

The investigators have developed a two-pronged approach (combining the FLASH technique and Guided Imagery) that aims to reduce existing symptoms of distress and provide participants with techniques to help them cope with future stressful events. This approach has been developed with experienced psychological practitioners, and staff members. The FLASH technique is a recently developed therapy which aims to reduce psychological distress following traumatic events. It allows participants to process traumatic memories without feeling distress. Using guided imagery, a trained psychological practitioner helps participants to direct attention from distressing or intrusive memories, by evoking or generating positive mental images, sounds, tastes, smells and movement. Emerging evidence suggests that both techniques are safe and effective.

PROACTIVE will investigate the feasibility and acceptability of this two-pronged approach to address existing traumatic symptoms and enhance future resilience for intensive care nurses. Findings will inform the design of a larger trial which tests intervention effectiveness.

DETAILED DESCRIPTION:
Nursing staff from critical care units within three Trusts will be approached, given information regarding the study, and invited to participate. Nurses who wish to take part will complete a consent form and a baseline range of psychological questionnaires. They will then be asked to join our group sessions; two guided imagery training sessions to enhance resilience; two therapy sessions, using the Flash Technique, to address symptoms of distress; and a final follow-up session to consolidate techniques learnt. Sessions will be delivered online, in four groups of ten staff. Recruitment will continue until the 40 intervention slots have been filled. Six months after the first intervention session, participants will be asked to repeat the range of psychological questionnaires, to help us understand whether the intervention helped to reduce psychological distress.

The investigators will report recruitment and adherence rates and collect preliminary data regarding the effectiveness of the intervention. The investigators will also undertake a process evaluation, to examine acceptability and give participants a chance to report their experience of the study.

Results will inform the design of a subsequent multi-centre trial investigating the effectiveness of the intervention in improving the mental wellbeing of intensive care nurses.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care nursing staff with experience of caring for critically ill patients with serious SARS-CoV2 infection

Exclusion Criteria:

* Currently receiving psychological support/treatment
* Pre-existing diagnosis of psychosis
* 'Reservist' nursing staff who were drafted in to look after ICU patients during the Covid-19 pandemic, but normally work elsewhere

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility 1 - Recruitment | 1 month post-recruitment end date
  Recruitment of at least 5 participants per month per site
Feasibility 2 - Protocol fidelity | 1 month post-intervention final session
  Adherence to >75% of protocol interventions
Feasibility 3 - Blinded outcome assessments | 6 months post-intervention
  Completed blinded outcome assessments in >75% of participants (by questionnaire). This will be calculated as a percentage of how many participants complete the questionnaire pack versus how many are enrolled on the trial.
Feasibility 4 - Participant retention | 6 months post-intervention
  Participant retention to study completion
Feasibility 5 - Acceptability of intervention | Between 6 and 12 months post-intervention
  Acceptability of intervention and assessments which will be assessed through the use of questionnaires and focus groups.

SECONDARY OUTCOMES:
Mental wellbeing | Baseline, 6 months post-intervention
  Warwick-Edinburgh Mental Wellbeing Scale - WEMWBS. Respondents rate items based on how often they have had the thought or feeling over the last two weeks, from 1 'not at all' to 5 'all of the time'. Total score is the sum of all items and ranges from 14-70. The higher the score, the higher the level of mental wellbeing.
Post-traumatic stress disorder | Baseline, 6 months post-intervention
  PTSD checklist - PCL-5. A 20 item self-report measure to assesses symptoms of PTSD over the last month. Items are rated on a 5-point scale ranging from 0 'not at all' to 4 'extremely'. Total score ranges from 0 to 80. A score of between 31-33 or above is indicative of probable PTSD.
Anxiety | Baseline, 6 months post-intervention
  Generalised Anxiety Disorder-7 - GAD-7. Items are rated for how often they have bothered the respondent over the last two weeks, from 0 'not at all' to 3 'nearly every day'. Total score is the sum of all items and ranges from 0 to 15. Scores of 5, 10, and 15 are the cut-off points for mild, moderate and severe anxiety, respectively.
Depression | Baseline, 6 months post-intervention
  Patient Health Questionnaire-9 - PHQ-9. This 9-item self-report measure assesses symptoms of depression. Items are rated for how often they have bothered the respondent over the last two weeks, from 0 'not at all' to 3 'nearly every day'. Total score is the sum of both items and ranges from 0 to 27. Depression severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Quality of life EQ-5D-5L | Baseline, 6 months post-intervention
  EuroQol Five Dimension- Five level scale - EQ-5D-5L. The 5-level version of the EuroQol-5D (EQ-5D-5L) is a brief measure for assessing general quality of life and health status. Items assess mobility, self-care, usual activities, pain/discomfort and anxiety/depression each on a 5-point scale. 5 items are scored on a 5-point ordinal scale from 'no problem' (1) to 'highest level of problems' (5). Respondents also rate their overall health today from 0 (the worst health you can imagine) to 100 (the best health you can imagine). Scores are analysed separately (not summed).
Resilience | Baseline, 6 months post-intervention
  Brief Resilience Scale - BRS. 6 items are scored on a 5-point ordinal scale from 'strongly disagree' to 'strongly agree', with reversing scores assigned to alternating questions. The scores for all 6 items are summed (giving a range from 6-30) and then divided by the total number of questions answered to give a final score.
Burnout syndrome | Baseline, 6 months post-intervention
  Maslach Burnout Inventory - MBI. 22 statements of job-related feelings for which respondents are asked the frequency to which they feel this way about their job ranging from 0 'never' to 6 'every day'. Each statement relates to one of three dimensions of burnout; emotional exhaustion, depersonalization and personal accomplishment. Each dimension is scored by summing the answer for that section and dividing by the number of items answered. Possible scores range as follows; EE 0-54, D 0-30 and PA 0-40, with a higher score associated with a higher level of burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Bates, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, United Kingdom